CLINICAL TRIAL: NCT03476135
Title: Immunogenicity and Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine Administered as a Booster Dose in Children Vaccinated 3 Years Earlier as Toddlers
Brief Title: Immunogenicity and Safety of a Booster Dose of a Quadrivalent Meningococcal Conjugate Vaccine in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MET62; 2017-001993-40 (EudraCT Number); U1111-1183-5988 (Other: WHO (Universal Trial Number))
Record Dates: First submitted 2018-03-19; First posted 2018-03-23 (Actual); Results first posted 2020-06-05 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Meningococcal Infections
Keywords: Meningococcal Meningitis; MenACYW conjugate vaccine; Quadrivalent meningococcal vaccine
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) (Experimental): Participants who received a single dose of MenACYW conjugate vaccine 3 years earlier in a previous vaccine study (MET54), received a booster dose of MenACYW conjugate vaccine at Day 0 in this study (MET62).
  Interventions: Biological: MenACYW conjugate vaccine
- Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix) (Experimental): Participants who received a single dose of Nimenrix® vaccine 3 years earlier in a previous vaccine study (MET54), received a booster dose of MenACYW conjugate vaccine at Day 0 in this study (MET62).
  Interventions: Biological: MenACYW conjugate vaccine

INTERVENTIONS:
Biological: MenACYW conjugate vaccine — Meningococcal polysaccharide (serogroups A, C, Y, and W) tetanus toxoid conjugate vaccine 0.5 mL, intramuscular

SUMMARY:
This was an open-label, multi-center study to describe the immune persistence of the priming dose and describe the immunogenicity and safety of a booster dose of Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid (MenACYW) conjugate vaccine in children in Finland who had been vaccinated 3 years earlier as toddlers with either MenACYW conjugate vaccine or Nimenrix® as part of the MET54 study (NCT03205358).

The objectives were:

* To describe the antibody persistence of meningococcal serogroups A, C, Y, and W before a booster dose in children who received either MenACYW conjugate vaccine or Nimenrix® 3 years earlier as toddlers.
* To describe the antibody responses to meningococcal serogroups A, C, Y, and W 30 days after a booster dose of MenACYW conjugate vaccine in children who received either MenACYW conjugate vaccine or Nimenrix® 3 years earlier as toddlers.
* To describe the antibody responses against tetanus toxoid 30 days after a booster dose of MenACYW conjugate vaccine in children who received either MenACYW conjugate vaccine or Nimenrix® 3 years earlier as toddlers.
* To describe the safety profile of a booster dose of MenACYW conjugate vaccine in children who received either MenACYW conjugate vaccine or Nimenrix® 3 years earlier as toddlers.

DETAILED DESCRIPTION:
Healthy children who were vaccinated 3 years earlier at 12 to 23 months of age in study MET54 (NCT03205358) were eligible for enrollment. All participants received a single booster dose of MenACYW conjugate vaccine on Day 0. Immunogenicity was assessed at pre-vaccination and 30 days after vaccination. Safety was assessed throughout the study period, and included solicited injection site and systemic reactions (Day 0 to Day 7 post-vaccination); unsolicited adverse events up to Day 30 (Visit 2), and serious adverse events occurring throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Participated in and completed (attended Visit 2) study MET54.
* Informed consent form had been signed and dated by the parent(s) or another legally acceptable representative (and by an independent witness, if required by local regulations).
* Participant and parent/legally acceptable representative were able to attend all scheduled visits and complied with all trial procedures.
* Covered by health insurance where applicable.

Exclusion Criteria:

* Participation in the 4 weeks preceding the trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks (28 days) preceding the trial vaccination or planned receipt of any vaccine prior to Visit 2 except for influenza vaccination, which might be received at a gap of at least 2 weeks before or after the study vaccines. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines. If the participant was due to receive vaccination(s) recommended for his/her age by the national immunization schedule at the time of the study, the participant was recommended to complete his/her immunization schedule after Visit 2.
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine (i.e., mono- or polyvalent, polysaccharide, or conjugate meningococcal vaccine containing serogroups A, C, Y, or W; or meningococcal B vaccine) with the exception of the single dose of meningococcal vaccine administered as part of study MET54.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* History of meningococcal infection, confirmed either clinically, serologically, or microbiologically
* At high risk for meningococcal infection during the trial (specifically, but not limited to, participants with persistent complement deficiency, with anatomic or functional asplenia, or participants traveling to countries with high endemic or epidemic disease).
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances.
* Verbal report of thrombocytopenia, contraindicating intramuscular vaccination in the Investigator's opinion.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination.
* Personal history of Guillain-Barré syndrome.
* Personal history of an Arthus-like reaction after vaccination with a tetanus toxoid-containing vaccine.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with trial conduct or completion.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature >= 38.0 degree Celsius [°C]). A prospective participant was not included in the study until the condition had resolved or the febrile event had subsided.
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw.
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study.

Ages: 46 Months to 61 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (8):
- Finland (8):
  - Sanofi Pasteur Investigational Site 2460005, Espoo
  - Sanofi Pasteur Investigational Site 2460006, Helsinki
  - Sanofi Pasteur Investigational Site 2460002, Helsinki
  - Sanofi Pasteur Investigational Site 2460007, Jarvenpaa
  - Sanofi Pasteur Investigational Site 2460008, Oulu
  - Sanofi Pasteur Investigational Site 2460001, Pori
  - Sanofi Pasteur Investigational Site 2460003, Tampere
  - Sanofi Pasteur Investigational Site 2460004, Turku

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 8 sites in Finland from 27 February 2018 to 10 September 2018.
Pre-assignment Details: A total of 91 participants who received a single dose of Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid (MenACYW) conjugate vaccine or Nimenrix® vaccine in previous study MET54 (NCT03205358) were enrolled in this study (MET62).
Period: Overall Study
Arm/Group | Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) | Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix)
Started | 42 | 49
Completed | 42 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) | Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix) | Total
Number analyzed (Participants) | 42 | 49 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.9 (0.35) | 3.9 (0.33) | 3.9 (0.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 30 | 46
  Male | 26 | 19 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Antibody Titers Measured by Serum Bactericidal Assay Using Human Complement (hSBA) Against Meningococcal Serogroups A, C, Y, and W Before a Booster Dose of MenACYW Conjugate Vaccine in MET62
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by hSBA.
Time Frame: Day 0 (pre-vaccination)
Population: Analysis was performed on Per-Protocol Analysis Set (PPAS) which included all participants who received at least 1 dose of the study vaccine, had a valid post-vaccination blood sample result and had no certain protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) | Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix)
Number analyzed (Participants) | 40 | 44
titers (1/dilution)
  Serogroup A | 12.1 [8.15 to 18.1] | 16.5 [11.9 to 22.9]
  Serogroup C | 106 [73.2 to 153] | 11.7 [7.03 to 19.4]
  Serogroup Y | 30.9 [24.2 to 39.5] | 17.6 [13.1 to 23.7]
  Serogroup W | 48.5 [34.4 to 68.4] | 21.9 [14.7 to 32.7]

2. Primary Outcome: Antibody Titers Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W After a Booster Dose of MenACYW Conjugate Vaccine in MET62
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by hSBA.
Time Frame: Day 30 (post-booster vaccination)
Population: Analysis was performed on PPAS.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) | Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix)
Number analyzed (Participants) | 40 | 44
titers (1/dilution)
  Serogroup A | 763 [521 to 1117] | 659 [427 to 1017]
  Serogroup C | 5894 [4325 to 8031] | 1592 [1165 to 2174]
  Serogroup Y | 2013 [1451 to 2792] | 2806 [2066 to 3813]
  Serogroup W | 2656 [1601 to 4406] | 3444 [2387 to 4970]

3. Primary Outcome: Antibody Titers Measured by Serum Bactericidal Assay Using Baby Rabbit Complement (rSBA) Against Meningococcal Serogroups A, C, Y, and W Before a Booster Dose of MenACYW Conjugate Vaccine in MET62
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by rSBA.
Time Frame: Day 0 (pre-vaccination)
Population: Analysis was performed on PPAS. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) | Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix)
Number analyzed (Participants) | 39 | 44
titers (1/dilution)
  Serogroup A | 135 [58.0 to 314] | 281 [131 to 606]
  Serogroup C | 102 [60.9 to 169] | 11.9 [6.14 to 22.9]
  Serogroup Y | 119 [65.0 to 219] | 126 [69.1 to 230]
  Serogroup W | 113 [54.6 to 234] | 126 [63.6 to 250]

4. Primary Outcome: Antibody Titers Measured by rSBA Against Meningococcal Serogroups A, C, Y, and W After a Booster Dose of MenACYW Conjugate Vaccine in MET62
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by rSBA.
Time Frame: Day 30 (post-booster vaccination)
Population: Analysis was performed on PPAS.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) | Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix)
Number analyzed (Participants) | 40 | 44
titers (1/dilution)
  Serogroup A | 4240 [3352 to 5365] | 5702 [4575 to 7107]
  Serogroup C | 8629 [6573 to 11328] | 4871 [3750 to 6327]
  Serogroup Y | 5499 [4502 to 6717] | 7814 [6465 to 9445]
  Serogroup W | 16103 [12691 to 20431] | 19793 [15538 to 25214]

5. Primary Outcome: Antibody Titers Measured by hSBA Against Meningococcal Serogroups A, C, Y, and W After Priming Vaccination in MET54 and Booster Vaccination in MET62
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by hSBA.
Time Frame: Day 0 (pre-vaccination) and Day 30 (post-priming vaccination) in study MET54, and Day 0 (pre-vaccination) and Day 30 (post-booster vaccination) in study MET62
Population: Analysis in both MET54 and MET62 was performed on Full Analysis Set for Persistence (FASP) which included all participants who had a valid pre-vaccination blood sample result. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) | Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix)
Number analyzed (Participants) | 42 | 49
titers (1/dilution)
  Serogroup A: Day 0 (MET54): number analyzed (Participants) | 41 | 49
  Serogroup A: Day 0 (MET54) | 3.68 [3.12 to 4.33] | 3.67 [3.15 to 4.29]
  Serogroup A: Day 30 (MET54) | 83.3 [63.9 to 109] | 49.6 [32.1 to 76.7]
  Serogroup A: Day 0 (MET62) | 11.9 [8.11 to 17.4] | 14.7 [10.7 to 20.2]
  Serogroup A: Day 30 (MET62): number analyzed (Participants) | 41 | 47
  Serogroup A: Day 30 (MET62) | 755 [520 to 1097] | 629 [418 to 948]
  Serogroup C: Day 0 (MET54) | 2.48 [2.04 to 3.01] | 2.30 [2.12 to 2.50]
  Serogroup C: Day 30 (MET54) | 594 [445 to 793] | 29.4 [20.1 to 43.1]
  Serogroup C: Day 0 (MET62) | 103 [71.7 to 149] | 11.6 [7.28 to 18.3]
  Serogroup C: Day 30 (MET62): number analyzed (Participants) | 41 | 47
  Serogroup C: Day 30 (MET62) | 5744 [4230 to 7800] | 1618 [1204 to 2172]
  Serogroup Y: Day 0 (MET54) | 2.17 [1.95 to 2.42] | 2.27 [2.05 to 2.52]
  Serogroup Y: Day 30 (MET54) | 105 [73.9 to 149] | 75.8 [54.2 to 106]
  Serogroup Y: Day 0 (MET62) | 32.5 [24.8 to 42.7] | 18.2 [13.8 to 24.0]
  Serogroup Y: Day 30 (MET62): number analyzed (Participants) | 41 | 47
  Serogroup Y: Day 30 (MET62) | 2048 [1486 to 2823] | 2710 [2022 to 3633]
  Serogroup W: Day 0 (MET54) | 2.00 [NA to NA] — The 95% confidence interval was not computable as the standard deviation of the sample was 0, since all participants had the same value. | 2.12 [2.00 to 2.24]
  Serogroup W: Day 30 (MET54) | 71.8 [53.3 to 96.7] | 40.1 [30.6 to 52.6]
  Serogroup W: Day 0 (MET62) | 50.0 [35.9 to 69.5] | 21.2 [14.6 to 30.9]
  Serogroup W: Day 30 (MET62): number analyzed (Participants) | 41 | 47
  Serogroup W: Day 30 (MET62) | 2776 [1682 to 4584] | 3235 [2278 to 4594]

6. Primary Outcome: Antibody Titers Measured by rSBA Against Meningococcal Serogroups A, C, Y, and W After Priming Vaccination in MET54 and Booster Vaccination in MET62
Description: Antibody titers against meningococcal serogroups A, C, Y, and W were measured by rSBA.
Time Frame: as for outcome 5
Population: Analysis in both MET54 and MET62 was performed on FASP. Here, 'Number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) | Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix)
Number analyzed (Participants) | 42 | 49
titers (1/dilution)
  Serogroup A: Day 0 (MET54) | 12.3 [5.25 to 28.8] | 4.88 [2.74 to 8.69]
  Serogroup A: Day 30 (MET54) | 3198 [2559 to 3996] | 7633 [5879 to 9909]
  Serogroup A: Day 0 (MET62): number analyzed (Participants) | 41 | 49
  Serogroup A: Day 0 (MET62) | 124 [54.0 to 283] | 239 [113 to 503]
  Serogroup A: Day 30 (MET62): number analyzed (Participants) | 41 | 47
  Serogroup A: Day 30 (MET62) | 4096 [3223 to 5205] | 5341 [4275 to 6674]
  Serogroup C: Day 0 (MET54) | 2.21 [1.81 to 2.70] | 2.15 [1.86 to 2.47]
  Serogroup C: Day 30 (MET54) | 2711 [2156 to 3409] | 414 [283 to 607]
  Serogroup C: Day 0 (MET62): number analyzed (Participants) | 41 | 49
  Serogroup C: Day 0 (MET62) | 94.4 [55.9 to 160] | 11.2 [6.11 to 20.6]
  Serogroup C: Day 30 (MET62): number analyzed (Participants) | 41 | 47
  Serogroup C: Day 30 (MET62) | 8474 [6483 to 11075] | 4817 [3759 to 6175]
  Serogroup Y: Day 0 (MET54) | 2.88 [1.87 to 4.42] | 4.29 [2.48 to 7.44]
  Serogroup Y: Day 30 (MET54) | 2667 [2063 to 3447] | 2836 [2127 to 3781]
  Serogroup Y: Day 0 (MET62): number analyzed (Participants) | 41 | 49
  Serogroup Y: Day 0 (MET62) | 120 [67.1 to 213] | 123 [67.6 to 223]
  Serogroup Y: Day 30 (MET62): number analyzed (Participants) | 41 | 47
  Serogroup Y: Day 30 (MET62) | 5553 [4565 to 6755] | 7498 [6213 to 9049]
  Serogroup W: Day 0 (MET54) | 2.00 [NA to NA] — The 95% confidence interval was not computable as the standard deviation of the sample was 0, since all participants had the same value. | 2.24 [1.78 to 2.81]
  Serogroup W: Day 30 (MET54) | 5793 [4346 to 7720] | 4214 [3162 to 5616]
  Serogroup W: Day 0 (MET62): number analyzed (Participants) | 41 | 49
  Serogroup W: Day 0 (MET62) | 106 [51.6 to 219] | 113 [57.9 to 219]
  Serogroup W: Day 30 (MET62): number analyzed (Participants) | 41 | 47
  Serogroup W: Day 30 (MET62) | 15839 [12530 to 20023] | 18710 [14737 to 23753]

7. Primary Outcome: Antibody Concentrations Against Tetanus Toxoid Before a Booster Dose of MenACYW Conjugate Vaccine in MET62
Description: Anti-tetanus antibodies were measured by electrochemiluminescent (ECL) assay.
Time Frame: Day 0 (pre-vaccination)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: International unit per milliliter(IU/mL)
Arm/Group | Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) | Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix)
Number analyzed (Participants) | 39 | 44
International unit per milliliter(IU/mL) | 3.12 [2.05 to 4.75] | 3.02 [2.11 to 4.31]

8. Primary Outcome: Antibody Concentrations Against Tetanus Toxoid After a Booster Dose of MenACYW Conjugate Vaccine in MET62
Description: Anti-tetanus antibodies were measured by ECL assay.
Time Frame: Day 30 (post-booster vaccination)
Population: Analysis was performed on PPAS.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) | Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix)
Number analyzed (Participants) | 40 | 44
IU/mL | 10.4 [8.41 to 12.8] | 9.36 [7.61 to 11.5]

9. Primary Outcome: Number of Participants With Immediate Adverse Event After Vaccination in MET62
Description: Immediate events captured medically relevant unsolicited systemic adverse events (AEs) that occurred within the first 30 minutes after vaccination. An unsolicited AE was an observed AE that did not fulfill the conditions pre-listed in the case report book (CRB) in terms of diagnosis and/or onset window post-vaccination. Systemic AEs were all AEs that were not injection or administration site reactions.
Time Frame: Within 30 minutes after vaccination
Population: Analysis was performed on safety analysis set which included participants who had received at least one dose of the study vaccine and had any safety data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) | Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix)
Number analyzed (Participants) | 42 | 49
Participants | 0 | 0

10. Primary Outcome: Number of Participants With Solicited Injection Site Reactions and Systemic Reactions in MET62
Description: A solicited reaction (SR) was an adverse reaction (AR) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRB. Solicited injection site reactions: pain, erythema, and swelling. Solicited systemic reactions: fever, headache, malaise and, myalgia.
Time Frame: Within 7 days after vaccination
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) | Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix)
Number analyzed (Participants) | 42 | 49
Participants
  Pain | 26 | 35
  Erythema | 22 | 27
  Swelling | 16 | 19
  Fever | 3 | 4
  Headache | 8 | 14
  Malaise | 13 | 15
  Myalgia | 14 | 21

11. Primary Outcome: Number of Participants With Unsolicited Adverse Event After Vaccination in MET62
Description: An unsolicited AE was an observed AE that did not fulfill the conditions pre-listed in the CRB in terms of diagnosis and/or onset window post-vaccination.
Time Frame: Within 30 days after vaccination
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) | Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix)
Number analyzed (Participants) | 42 | 49
Participants | 22 | 15

12. Primary Outcome: Number of Participants With a Serious Adverse Event (SAE) After Vaccination in MET62
Description: A SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was an important medical event.
Time Frame: Within 30 days after vaccination
Population: Analysis was performed on safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) | Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix)
Number analyzed (Participants) | 42 | 49
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: SR were collected up to Day 7 after each vaccination, non-serious unsolicited AEs were collected up to Day 30 after each vaccination. SAEs were collected throughout the trial (up to 30 days after vaccination).
Description: SR was an AR observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRB. An unsolicited AE was an observed AE that did not fulfill the conditions pre-listed in the CRB in terms of diagnosis and/or onset window post-vaccination. Analysis was performed on safety analysis set.
Arm/Group | Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) | Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/49
Other Adverse Events (participants affected / at risk) | 36/42 | 43/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1:MenACYW Conjugate Vaccine(Previous Exposed to MenACYW) (N=42) | Group2:MenACYW Conjugate Vaccine(Previous Exposed to Nimenrix) (N=49)
Injection Site Erythema (General disorders) | 22 (22) | 27 (27)
Injection Site Pain (General disorders) | 26 (26) | 35 (35)
Injection Site Swelling (General disorders) | 16 (16) | 19 (19)
Malaise (General disorders) | 13 (13) | 15 (15)
Pyrexia (General disorders) | 3 (3) | 4 (4)
Otitis Media (Infections and infestations) | 1 (1) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 7 (7) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 14 (14) | 21 (21)
Headache (Nervous system disorders) | 10 (11) | 14 (14) — Headache events that occurred after 7 days post-vaccination were considered as unsolicited AE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2018-03-15): https://cdn.clinicaltrials.gov/large-docs/35/NCT03476135/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT03476135/SAP_001.pdf